CLINICAL TRIAL: NCT06500871
Title: Evaluation of the Effect of Intra-ligamentary Injection of Diclofenac Potassium Versus Articaine on Anaesthetic Efficacy in Mandibular Molars With Symptomatic Irreversible Pulpitis:A Randomized Controlled Trial
Brief Title: Evaluation of the Effect of Intra-ligamentary Injection of Diclofenac Potassium Versus Articaine on Anaesthetic Efficacy in Mandibular Molars With Symptomatic Irreversible Pulpitis.
Status: Not yet recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mai Abdou Ibraheem, Resident at faculty of dentistry, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ENDO 9-1-2
Record Dates: First submitted 2024-07-08; First posted 2024-07-15 (Actual); Last update posted 2024-08-06 (Actual); Status verified 2024-08

CONDITIONS: Teeth With Acute Irreverseble Pulpitis
MeSH Terms: interventions — Diclofenac

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Diclofenac Potassium (Experimental): 0.4 ml diclofena potassium injection 75mg/3ml drug used as Supplemental intraligamentary injection
  Interventions: Drug: Diclofenac Potassium
- Articaine Anaesthetic solution (Active Comparator): Articaine 4% with (1:100,000 Epinephrine) local anesthetic solution will be used as intraligamentary injection,
  Interventions: Drug: Diclofenac Potassium

INTERVENTIONS:
Drug: Diclofenac Potassium — NSAID

SUMMARY:
This study aims to assess the effect the intraligamentary injection of Diclofenac Potassium versus Articaine 4% on the anaesthetic efficacy & intensity of intraoperative & postoperative pain during single visit root canal treatment in patients with symptomatic irreversible pulpitis in mandibular molar teeth

ELIGIBILITY:
Inclusion Criteria:

* Systemically healthy patient (ASA I or II).
* Mandibular Posterior teeth with:

Preoperative sharp pain, Absence or slight widening in the periodontal ligament (PDL), Vital response of pulp tissue to cold pulp test.

* patients who agree to provide written consent and the patients able to understand the pain scale and attend for recall appointments

Exclusion Criteria:

1. Patients allergic to anesthetic solutions & other NSAIDs.
2. Pregnant or nursing females.
3. Patients having significant systemic disorder (ASA III or IV).
4. Gastrointestinal disorders.
5. If the initial diagnosis revealed pain in more than one tooth.
6. Hemostatic disorders or anti-coagulant therapy during the last month.
7. Consumption of opioid or non-opioid analgesics or NSAIDs during the last 12 hours before treatment.
8. Teeth that have:

   i. Periodontal involvement (with pocket depth greater than 5mm, associated with swelling or fistulous tract, or greater than grade I mobility).

   ii. No possible restorability. iii.Signs of pulpal necrosis; associated sinus tract or swelling.

   -

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-08 (Estimated); Primary Completion 2025-05 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
Efficacy of local anesthesia | intraoperative ( access cavity preparation & instrumentation ) during root canal treatment
  using Heft parker Visual Analogue scale Binary where success is defined as no pain or faint/weak /mild pain<55 mm). if >55 defined as failure

SECONDARY OUTCOMES:
Intensity of intraoperative pain | intraoperative ( access cavity preparation & instrumentation ) during root canal treatment
  using Heft parker Visual analogue scale score ranges from on a 170-mm VAS line with the ends labeled "no pain" and "unbearable pain. .no pain (< 5 mm), mild pain (≥ 5 mm and ≤ 54 mm), Moderate pain (> 54 mm and < 114 mm), Severe pain (≥ 114 mm).
Post-operative pain | 6, 12, 24 and 48 hours post-operatively
  using Heft parker Visual analogue scale on a 170-mm VAS line with the ends labeled "no pain" and "unbearable pain. .no pain (< 5 mm), mild pain (≥ 5 mm and ≤ 54 mm), Moderate pain (> 54 mm and < 114 mm), Severe pain (≥ 114 mm).
Number of needed analgesic tablets in case of intolerable pain | Up to 2 days post operatively
  by counting